CLINICAL TRIAL: NCT05869812
Title: Influence of β-hydroxy β-methyl Butyrate (HMB)Supplementation on Post-operative Muscle Mass and Function in Female Athletes
Acronym: FAKS-HMB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Strength and Conditioning Association (Other); Metabolic Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Ashley A. Herda, Ph.D., CSCS*D, Assistant Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00149057
Record Dates: First submitted 2023-03-14; First posted 2023-05-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atrophy
Keywords: musculoskeletal
MeSH Terms: conditions — Atrophy | interventions — Dietary Supplements; beta-hydroxyisovaleric acid; calcium lactate

STUDY DESIGN:
Intervention Model Description: This study will be conducted in a randomized, double-blind, placebo-controlled clinical trial where practitioners and participants will be blinded to the supplementation treatment (experimental product versus placebo control)
Who Masked: Participant, Investigator
Masking Description: The sponsor- investigator, Dr. Ashley Herda, will provide the participants with the investigational product or placebo in identical, yet coded product containers and the product manufacturer, MTI BioTech, Inc., will retain the blind code until completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CaHMB+Vitamin D3-Active Experimental (Experimental): Participants will consume 3 g HMB with 2000 IU Vitamin D3 per day, split into two doses daily for the duration of the study, beginning 2 weeks prior to their surgical date. The first dose will be consumed 60 minutes prior to any at- home or outpatient physical therapy session and a second will be consumed immediately following the session. If a treatment day does not include any rehabilitation session, the participant will consume one dose in the morning prior to food consumption and the second dose approximately 90 minutes later.
  Interventions: Drug: CaHMB (Dietary supplement, not Drug)
- Calcium Lactate-Control Placebo (Placebo Comparator): Participants will consume inactive 510 mg Ca Lactate capsules per day, split into two doses daily for the duration of the study, beginning 2 weeks prior to their surgical date. The first dose will be consumed 60 minutes prior to any at- home or outpatient physical therapy session and a second will be consumed immediately following the session. If a treatment day does not include any rehabilitation session, the participant will consume one dose in the morning prior to food consumption and the second dose approximately 90 minutes later.
  Interventions: Dietary Supplement: CaLa

INTERVENTIONS:
Drug: CaHMB (Dietary supplement, not Drug) — The investigators will focus our effort, for the purposes of this study, on determining if adding an HMB supplement will stimulate positive outcomes and recovery of the quadriceps and hamstrings muscle architecture and function in females with ACL injury requiring surgical repair, more so than a placebo control.
  Other Names: Calcium HMB; Beta-hydroxy-beta-methylbutyrate
  Arms: CaHMB+Vitamin D3-Active Experimental
Dietary Supplement: CaLa — Comparative placebo
  Other Names: Calcium Lactate
  Arms: Calcium Lactate-Control Placebo

SUMMARY:
The proposed project will evaluate the musculoskeletal outcomes of quadriceps and hamstring muscle size and function following orthopedic knee surgery involving anterior cruciate ligament (ACL) repair or reconstruction. Currently, the research team collaborates with a team of orthopedic specialists at the University of Kansas Health System and monitor muscle size post-knee repair and follow the standard of care (SOC) practices of the licensed physical therapists (PT). The proposed project will include a randomized clinical trial to observe the muscular outcomes following the current SOC plus supplementation of calcium-β-hydroxy-β-methylbutyrate (caHMB) or placebo. CaHMB has been shown to improve rates of muscle protein synthesis while suppressing muscle protein breakdown in healthy adults. The use of caHMB has also provided evidence of muscular protection from atrophy during prolonged bed rest. This evidence supports the utility in clinically injured athletes that are subjected to disuse atrophy from the inability to bear weight or participate in typical daily physical activity. Additionally, matched for activity-related knee injuries, female athletes are more susceptible to incurring a significant injury due to a variety of genetic, hormonal, biological, anatomical, and biomechanical predispositions. Therefore, the proposed study will recruit approximately 30 females over the age of 18 that have sustained an injury to the ACL and will plan to undergo reconstructive knee surgery involving the ACL. Subjects will be monitored and measured prior to their surgical date (T0), at 2-weeks post operative (T1), and every 6-weeks until they are cleared to return to sport (T2-TRTS). Participants will be randomly assigned 1:1 in a double-blind manner to either an experimental (EXPHMB) or placebo (CONPLA) group. Doses will be provided to the participants in coded containers and will complete their dosing and a record log of intake for the duration of their rehabilitation. Three 3-day food, exercise, and health record logs will be collected to monitor nutritional intake, activity, and menstrual patterns at T0, T3, and TRTS. Participant's assessments will include body composition analysis via bioelectrical impedance analysis for total and segmental muscle and fat mass, skeletal muscle mass, and body fat percent. We will collect ultrasound images of the quadriceps and hamstrings of the operative-involved limb (OPIL) and non-operative limb (NOPL) limbs for muscle cross-sectional area (mCSA), thickness (mT), subcutaneous fat thickness (TFAT), and corrected echo intensity (EICOR) at all time points. Strength and functional assessments will occur upon entrance to the study (T0), and after loaded exercise is indicated by the practitioner (T3-TRTS) to the tolerance of the athlete. These assessments include maximal voluntary isometric contractions (MVIC) for leg extension and leg curl, standing balance tests, single-leg and double-leg jump assessment, and drop landing deviation, all on dual force plates. Data will be analyzed using multiple three-way analyses of variance [surgical leg (OPIL vs. NOPL) x treatment (EXPHMB vs. CONPLA) x time (T0 vs. T1 vs. T2 vs. T3 vs. T4 vs. T5 vs. TRTS) for the dependent variables. Significance is established at p≤0.05 and follow-up ANOVAS, T-tests, and post-hoc analyses will be conducted when significance is present. The evidence from this study will support the practitioners and coaches' abilities to maximize recovery and training outcomes, respectively, in previously injured female athletes.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written and dated informed consent to participate in the study.
2. Participant is biological female between 18 and 45 years of age, inclusive.
3. Participant intends to complete postoperative rehabilitation at affiliated physical therapy clinic.

Exclusion Criteria:

1. Participant is currently consuming nutritional supplements or has recently (regularly) consumed nutritional supplements, other than multivitamins and minerals in <9 weeks prior to participation.
2. Participant currently suffers from a sleep disorder and/or has a known history of (or is currently being treated for) clinical depression, eating disorder(s) or any other psychiatric condition(s) that might limit natural recovery from substantial injury.
3. Participant has a history of orthopedic injury or surgery within the last year in the non-operative limb that may prevent them from completing the study procedures.
4. Participant has history of previous injury or surgery in the operative limb.
5. Participant has implants, hardware, devices, or other non-removable metal material in the body that would limit the accuracy of body composition assessments within the measurement area.
6. Participant is participating in another clinical trial or has received an investigational product within thirty days prior to enrollment.
7. Participant has a known allergy or sensitivity to any ingredient in the test product/s.
8. Participant is pregnant as confirmed by a urine sample and hCG test.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in leg lean muscle mass | every 6 weeks for 9-months
  absolute leg lean mass (kg) change from baseline
Change in leg lean muscle mass | every 6 weeks for 9-months
  absolute muscle cross-sectional area (cm^2)
Muscle Mass | every 6 weeks for 9-months
  percent change cross-sectional area (%)

SECONDARY OUTCOMES:
Isometric leg strength change | every 3 months for 9-months
  change in strength from baseline relative to contralateral limb (kg)
Change in EMG amplitude | every 3 months for 9-months
  absolute (RMS) change from baseline

OTHER OUTCOMES:
ALM body composition change | every 6 weeks for 9-months
  appendicular lean mass (kg) change from baseline
Fat mass body composition change | every 6 weeks for 9-months
  fat mass (kg) change from baseline
TBLM body composition change | every 6 weeks for 9-months
  total body lean mass (kg) change from baseline
Functional performance Asymmetry Index | measured at 14 and 26 weeks
  symmetry difference between limbs, expressed as a percent Drop landing knee excursion (force, impulse) Vertical jump (height, force, impulse) Cross-over hop (distance) Single-leg hop (distance) Triple hop (distance) Figure-8 hop (time-sec.) Number of leg press repetitions
  All scores aggregate to a single percent score comparing operative limb to non-operative limb.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Health System, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No